CLINICAL TRIAL: NCT04869774
Title: A Mobile Application for Wound and Symptom Surveillance After Colorectal Surgery: a Feasibility Randomized Controlled Trial
Brief Title: Wound And Symptom Tracking After Colorectal Surgery Using How2trak
Acronym: WATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ottawa (Other)
Collaborators: The Ottawa Hospital (Other); Health Outcomes Worldwide (Unknown)
Responsible Party: Principal Investigator, Reilly Patrick Musselman, Principal Investigator, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20200596-01H
Record Dates: First submitted 2021-04-23; First posted 2021-05-03 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Surgical Site Infection; Mobile Applications; Surgery--Complications; Colorectal Surgery
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Masking Description: This study will be unblinded so no attempts at concealment of individuals' allocation will be made.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Monitoring (Active Comparator): Patients discharged from hospital after colorectal surgery will have virtual monitoring of their surgical incision and symptoms, using the mobile application How2Trak, post-operatively.
  Interventions: Device: How2Trak mobile application
- Standard of Care (No Intervention): Patients discharged from hospital after colorectal surgery will receive standard of care with no virtual monitoring of their surgical incision and symptoms.

INTERVENTIONS:
Device: How2Trak mobile application — Patients will undergo virtual monitoring of their incision and symptoms using the How2Trak application(app). Using the app, patients will be asked to answer a series of questions and photograph their surgical incision on post-operative day 3, 5, 7, 10, 20, and 30. Patient responses and photographs entered into the app will be reviewed within 72 hours by a trained Nurse Specialized in Wound, Ostomy and Continence. If a concern is identified the nurse will contact the patient to arrange a virtual visit using the how2trak app or notify the surgeon team (including colorectal surgeons and physician residents) in accordance with clinical discretion.
  Arms: Virtual Monitoring

SUMMARY:
The purpose of this study is to assess the feasibility of using a mobile application (app) called how2trak to improve people's experience, wound surveillance, and detection of surgical site infections (SSI) after colorectal surgery while reducing in-person interactions for patients during the COVID-19 pandemic.

This will inform the implementation of a full-scale trial to establish if surveillance of someone's incision and symptoms using how2trak improves SSI detection and management compared to standard care (involving a single post-operative surgery clinic visit).

The data collected will contribute to a broader dataset of people with SSI surveillance to be used in developing a clinical decision support system.

DETAILED DESCRIPTION:
Background: Surgical site infections (SSI) are the most common nosocomial infection and occur in 16.3% of individuals undergoing colorectal surgery at our institution, the majority of which are identified after discharge from hospital. Patients concerned to have an SSI, generally present to the emergency department or surgery clinic. Both options for in-person interaction are costly to the healthcare system and patients, and increase their risk of COVID-19 exposure. A mobile application How2trak has proven to be beneficial for patients with complex wounds at our institution by facilitating at-home monitoring and virtual consultations.

Aim: This study aims to assess the feasibility of a randomized controlled trial to assess if How2trak can improve patients' experience, and detection of surgical site infections after colorectal surgery while reducing their risk of COVID-19 exposure.

Methods: In this single-center, prospective feasibility trial, eligible patients undergoing elective and semi-urgent colorectal surgery will be randomized to either standard care or How2trak post-operative monitoring of their incision, symptoms, and ostomy function. Patient self-assessments will be monitored by a nurse specialized in wound and ostomy care who will meet virtually with the patient as needed. The primary outcome is feasibility as measured by enrollment, randomization, H2T usability, data extraction, and resource capacity.

Results: We anticipate this work will help us to better understand the feasibility of using mobile technology to optimize patients' care after discharge from hospital after colorectal surgery. Virtual post-surgery wound and symptom monitoring could enhance patient experience, SSI detection, and reduce the risk of COVID-19 transmission. If this technology is feasible for our patient population and workflow, next steps will be to assess its effectiveness with a full-scale randomized controlled trial and explore additional applications including ostomy monitoring, patient education, and application in other surgical departments.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 16 years of age or older who are being discharged from hospital after undergoing semi-urgent, urgent, or elective abdominal surgery by a colorectal surgeon at The Ottawa Hospital, and have provided informed consent to participate.

Patients enrolled in other clinical trials will still be candidates for this feasibility trial.

Clinicians using the how2trak app in this study will be considered study participants as well. They will be asked to complete the "Patient and Clinician Survey of Application". This survey addresses the experience with the use of the H2T app their feedback regarding usability is fundamental for future improvement.

Exclusion Criteria:

* Individuals will be excluded if less than 16 years of age; have no access or ability to use a mobile device; no cellular data/WiFi access; and/or cannot read and write in English.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Capability for enrollment | 6 months
  number of patients per month on average are enrolled in the study
Feasibility of the randomization processes | 6 months
  proportion of patients randomized to the intervention or control group.
How2trak compliance | 6 months
  Proportion of self-assessments completed by patients, on average.
How2trak usability, delivery and compliance | 6 months
  The mean score for the patient and clinician survey of H2T application.
Monitoring of protocol deviation and safety | 6 months
  The number and frequency of events when study activities diverge from the REB-approved protocol or are considered adverse events.
Feasibility of data extraction | 6 months
  Proportion of patients for which all primary outcomes of the definitive trial are recorded. This includes the SSI incidence and severity and patient experience.
Resources and time required to conduct the feasibility trial will be assessed | 8 months
  There is adequate administrative capacity, expertise, skills, space and time of the research team to complete the study.

SECONDARY OUTCOMES:
Surgical Site Infection (SSI) Rate | 6 months
  Secondary outcomes will include SSI incidence and severity.
Patient experience | 6 months
  Response to patient experience survey
Healthcare System Time | 6 months
  Hours of in-person interactions with the healthcare system, including readmissions to hospital, ED visits, clinic visits etc.
Covid-19 infection Rate | 6 months
  Confirmed COVID-19 infection within 30 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Reilly Musselman, MD, MSc, Principal Investigator — University of Ottawa; Heather Smith, MD, MSc, Principal Investigator — University of Ottawa

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD with other partners, collaborators, or researchers.
  Data will be captured through the assessments and/or photographs in the app and EPIC. Data sent from how2trak to TOH will be transferred through a secure, access-controlled folder within Office 365 including patient identifiers to allow for merging with EPIC data. Once the data files are merged, they will be deidentified. Only research personnel will have access to the study data. A data monitoring committee will not be developed given the minimal risk and small sample size of this feasibility trial.

REFERENCES:
- [Derived] Valk HA, Garcia-Ochoa C, Fontaine Calder J, Miller T, Rashidi B, McIsaac C, Musselman R. A Mobile App for Wound and Symptom Surveillance After Colorectal Surgery: Protocol for a Feasibility Randomized Controlled Trial. JMIR Res Protoc. 2022 Jan 14;11(1):e26717. doi: 10.2196/26717. PMID 34854816